CLINICAL TRIAL: NCT06514118
Title: Chemoimmunotherapy Plus Ratiotherapy for Extensive Stage Small-cell Lung Cancer
Brief Title: Chemoimmunotherapy Plus Residual Lesion Irradiation for the Treatment of Extensive Stage Small-cell Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: Qingdao Central Hospital (Other)
Responsible Party: Principal Investigator, Youxin Ji, Director, Qingdao Central Hospital
Other Study IDs: KY202400902
Record Dates: First submitted 2024-07-04; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Small-cell Lung Cancer; Residual Tumor; Radiation
MeSH Terms: conditions — Small Cell Lung Carcinoma; Neoplasm, Residual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Combined chemotherapy and immunotherapy plus residual lesion irradiation: Patients receive carboplatin 5/AUC intravenously (IV) on day 1, adebrelimab 1200mg IV on day 1, and etoposide100mg/m2 IV on days 1-3. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity; redsidual tumor irradiation for 50GY in 25 fraction.
  Interventions: Radiation: residual tumor irradiation

INTERVENTIONS:
Radiation: residual tumor irradiation — lung residual tumor will be given external beam irradiation for 50GY in 25 fractions in total

SUMMARY:
This is a phase II trial studies the effect of chemoimmunotherapy sequential residual tumor irradiation in treating patients with extensive stage small cell lung cancer. Even though small cell lung cancer is initially highly responsive to first-line chemotherapy plus PD-L1 inhibitors, treatment resistance inevitably happens. Residual tumor irradiation my prolong drug resistance, and may help prevent the growth and spread of the tumor cells to other parts of the body.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the progression-free survival (PFS) and overall survival of chemoimmunotherapy sequential residual tumor irradiation in patients with extensive stage small cell lung cancer (SCLC).

SECONDARY OBJECTIVES:

II. To assess the overall response rate (ORR) and toxicity in extensive stage SCLC patients treated with chemoimmunotherapy squential residual tumor irradiation

ELIGIBILITY:
Inclusion Criteria:

>= 18 years of age Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 1 at the time of study treatment initiation Histologically or cytologically confirmed diagnosis of small cell lung cancer (SCLC) Patient should have extensive stage disease, defined as, malignant pleural effusion, pulmonary metastases in the contralateral lung, and/or the presence of extra-thoracic metastatic disease Must have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 prior to starting platinum-based systemic chemotherapy Absolute neutrophil count (ANC) >= 1.5 x 10^9/L Platelets >= 100 x 10^9/L Hemoglobin >= 9 g/dL Serum creatinine =< 1.5 x institution upper limit of normal (ULN) and calculated creatinine clearance of at least 15 ml/min.

Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x upper limit of normal (ULN) (ALT and AST =< 5 x ULN is acceptable if liver metastases are present) Total serum bilirubin =< 1.5 x ULN. For patients with well documented Gilbert's syndrome, total bilirubin =< 3 x ULN with direct bilirubin within normal range.

Participant must understand the investigational nature of this study and sign an approved written informed consent form prior to receiving any study related procedure.

Exclusion Criteria:

* ad major surgery within 14 days prior to starting study drug or has not recovered from major side effects (tumor biopsy is not considered major surgery) resulting from a prior surgery Positive for immunosuppressive disease, acquired immunodeficiency syndrome (AIDS) or other immune depressing diseases. For human immunodeficiency virus (HIV), HVC and HBC-mandatory testing is required prior to enrollment Patient has known hypersensitivity to the components of the study drugs or any analogs History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, including, but not limited to: Myocardial infarction or arterial or venous thromboembolic events within 6 months prior to baseline or severe or unstable angina, New York Heart Association (NYHA) class III or IV disease. History of documented congestive heart failure (New York Heart Association functional classification III or IV) within 6 months prior to baseline. Poorly controlled arrhythmias

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with extensive disease of small-cell lung cancer are enrolled and treated with chemotherapy plus PD-L1 immunotherapy for 4 cycles. Patients with esponse or stable disease are selected to receive residual lesions irratiation for 50GY/25f.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2026-03-16 (Estimated); Study Completion 2027-03-16 (Estimated)

PRIMARY OUTCOMES:
progression-free survival (PFS) | 24 months
  PFS: time to disease progression or patient death

SECONDARY OUTCOMES:
Overall survival (OS) | 36 months
  OS: time to patient death

CONTACTS AND LOCATIONS:
Overall Officials: chunling zhang, md, Study Chair — Qingdao Central Hospital
Locations (1):
- Qingdao Central Hospital, Qingdao, Shandong, China